CLINICAL TRIAL: NCT07242313
Title: Comparative Study Between Demineralized and Mineralized Allogeneic Dentin Grafts for Alveolar Ridge Preservation: A Randomized Controlled Clinical Trial
Brief Title: Comparison of Demineralized and Mineralized Dentin Grafts in Ridge Preservation
Acronym: DDG-ARP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Abdelhamid Musa Abdelaziz, Master's Student, Department of Periodontology, Faculty of Dentistry, Kafrelsheikh University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KFSIRB200-718
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Alveolar Ridge Preservation; Post Extraction Alveolar Bone Resorption
Keywords: Alveolar Ridge Preservation; Socket Preservation; Post-Extraction Bone Loss; Dentin Graft; Allogeneic Dentin; Demineralized Dentin Matrix; Mineralized Dentin Graft; Bone Regeneration; Histomorphometry

STUDY DESIGN:
Intervention Model Description: Three-arm parallel-group randomized clinical trial comparing two types of allogeneic dentin grafts with a control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, outcome assessors, and the statistician are blinded to group allocation. Care providers are blinded to graft type in the demineralized and mineralized groups but not in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Demineralized Allogeneic Dentin Graft (Experimental): After atraumatic tooth extraction, the socket is filled with demineralized allogeneic dentin particulate graft. The material is processed and sterilized according to standardized laboratory protocols. A resorbable collagen dressing is placed over the graft, followed by site closure. This arm evaluates the regenerative effectiveness of demineralized dentin on ridge preservation.
  Interventions: Biological: Demineralized Allogeneic Dentin Graft
- Mineralized Allogeneic Dentin Graft (Experimental): Following atraumatic extraction, the socket is grafted with mineralized allogeneic dentin particulate material processed and sterilized under controlled conditions. A resorbable collagen dressing is applied prior to closure. This arm assesses the ridge preservation outcomes produced by the mineralized form of dentin graft.
  Interventions: Biological: Mineralized Allogeneic Dentin Graft
- Control: Spontaneous Healing (Empty Socket) (No Intervention): Participants in this arm undergo atraumatic tooth extraction followed by natural socket healing without graft placement. The socket is allowed to heal spontaneously to serve as the control for evaluating dimensional bone changes relative to grafted groups.

INTERVENTIONS:
Biological: Demineralized Allogeneic Dentin Graft — Particulate demineralized allogeneic dentin processed from donor teeth using standardized laboratory protocols, including cleaning, defatting, demineralization, dehydration, freeze-drying, and sterilization. The graft is placed into the extraction socket following atraumatic extraction, covered with a resorbable collagen dressing, and the site is closed to promote alveolar ridge preservation.
  Arms: Demineralized Allogeneic Dentin Graft
Biological: Mineralized Allogeneic Dentin Graft — Particulate mineralized allogeneic dentin derived from processed donor teeth. The dentin is cleaned, defatted, ultrasonically treated, dehydrated, freeze-dried, and sterilized while retaining its mineral phase. The graft is inserted into the extraction socket after atraumatic extraction and covered with a resorbable collagen material prior to closure to support ridge preservation.
  Arms: Mineralized Allogeneic Dentin Graft

SUMMARY:
This clinical investigation aims to assess how two different allogeneic dentin graft materials - one de-mineralized and the other mineralized - influence bone preservation following extraction of a single upper posterior tooth. A total of 45 patients will be randomly allocated into three equal groups: a socket-only spontaneous healing group (control), a de-mineralized dentin graft group, and a mineralized dentin graft group. Over a six-month period after extraction, measurements will be taken using CBCT to monitor changes in ridge width, height, and bone density. Secondary outcomes include patient-reported pain, postoperative swelling, satisfaction levels, width of keratinized tissue, and histomorphometric data from biopsy samples at implant placement. Findings from this trial may support evidence-based decisions in alveolar ridge preservation and help clinicians choose the most predictable grafting strategy before implant placement.

DETAILED DESCRIPTION:
The alveolar ridge experiences rapid remodeling after tooth extraction, often resulting in significant bone loss if no graft is placed. Clinical observations indicate that an extraction site may lose roughly half of its original width within six to twelve months, severely reducing the bone available for future implants or prosthetic support. This resorption occurs because removal of the tooth and its periodontal ligament eliminates the normal mechanical stimulation that maintains the surrounding bone. Alveolar ridge preservation techniques aim to counteract this remodeling by placing a graft in the extraction socket to maintain bone dimensions and support healing. Preserving the ridge anatomy in this way is critical for subsequent restorative procedures such as dental implant placement or denture support.

In practice, a variety of graft materials have been used to support alveolar ridge preservation. Autogenous bone grafts (harvested from the patient's own body, for example from the iliac crest or intraoral sites) have osteogenic and osteoinductive properties, but require a second surgical site and provide limited graft volume. Alternative materials include allogeneic bone (processed human bone from donors) and xenogeneic bone (such as bovine-derived hydroxyapatite), which are readily available but may integrate more slowly and raise concerns about immune reaction or disease transmission. Synthetic or alloplastic graft materials (calcium phosphates, bioactive glasses, polymers, etc.) are also used, although they typically act only as osteoconductive scaffolds and may not match the biologic activity of natural tissues. Given these limitations, there is ongoing interest in novel graft sources that can offer both safety and biological efficacy.

One promising graft material is dentin, the calcified tissue comprising the bulk of a tooth beneath the enamel. Chemically, dentin closely resembles bone: it is roughly 70% mineral (hydroxyapatite) and 20% organic matrix (predominantly type I collagen) by weight, along with non-collagenous proteins and embedded growth factors. Because dentin is acellular and avascular, it is inherently well-tolerated when used as a graft. Importantly, its organic matrix contains signaling molecules such as bone morphogenetic proteins (BMPs) and other growth factors that are naturally osteoinductive. In clinical practice, an extracted tooth can be cleaned and converted into graft material by grinding it into particulate form or shaping it into a block. Clinical studies have shown that autogenous tooth-derived grafts (using a patient's own extracted tooth) can effectively support socket preservation and guided bone regeneration. However, this approach is limited by the availability of teeth in each patient and by variability in processing methods, which can affect the consistency of the graft material.

Dentin grafts can be prepared in different forms. Demineralized dentin matrix (DDM) is produced by treating the dentin with acid to remove most of the mineral phase, leaving a collagen-rich matrix that retains the dentin's organic proteins and growth factors. DDM is highly osteoinductive: by removing the crystalline mineral, the embedded signaling molecules (such as BMPs and transforming growth factors) are exposed, creating a bioactive scaffold that strongly stimulates new bone formation. In contrast, a fully mineralized dentin graft (for example, ground whole tooth particles that are not demineralized) retains the hydroxyapatite content, which contributes rigidity and initial volume stability. These mineralized grafts act primarily as an osteoconductive scaffold and release bioactive molecules more slowly as they resorb. In practical terms, demineralized dentin grafts are believed to accelerate early bone ingrowth, whereas mineralized dentin grafts may better preserve the initial socket architecture and support gradual long-term remodeling.

Allogeneic dentin grafts are obtained from healthy human donor teeth that have been processed and sterilized under controlled conditions. The use of donated extracted teeth provides a scalable graft source and repurposes material that would otherwise be discarded. Processing typically involves cleaning away any attached soft tissues, removing enamel and cementum, and grinding the remaining tooth structure into particles. Sterilization (for example by freeze-drying, gamma irradiation, or other validated methods) ensures the graft is safe for implantation. For demineralized allografts, an additional acid step is applied to decalcify the particles. These preparation steps remove or inactivate cells and pathogens, minimizing immunogenic components. Preclinical studies suggest that properly processed allogeneic dentin matrix can induce bone formation with minimal immune reaction or rejection. However, standardized clinical evidence on allogeneic dentin grafts remains limited.

Given this background, the current trial is designed to determine which graft preparation yields better ridge preservation outcomes. Both demineralized and mineralized allogeneic dentin grafts are expected to support bone healing, but they may influence the process differently. Demineralized allogeneic dentin grafts, with their exposed collagen matrix and retained growth factors, may encourage rapid initial bone ingrowth. Mineralized allogeneic dentin grafts may offer greater immediate structural support and preserve socket volume over time, although they tend to release growth factors more slowly. The comparative performance of these two graft types in humans has not been established, creating a clear need for a controlled clinical study.

This randomized controlled clinical trial will enroll patients undergoing single-tooth extraction who require ridge preservation. Patients will be randomly assigned to receive either a demineralized allogeneic dentin graft or a mineralized allogeneic dentin graft placed into the fresh extraction socket. In each case the graft material will be placed immediately after extraction and the site will be closed using standard surgical technique. Both groups will follow the same postoperative care and follow-up protocol. After a predetermined healing interval (for example, three to six months), the sites will be re-entered for evaluation. Assessment will include clinical inspection and radiographic imaging of the ridge, and if feasible histological analysis of any newly formed bone, to compare bone volume and architecture between the two graft types.

This study addresses a gap in current clinical evidence, as no published trials have directly compared demineralized and mineralized human dentin grafts for socket preservation. Prior research has shown that autologous tooth-derived grafts can be effective for ridge preservation, but the optimal approach for donated (allogeneic) dentin remains uncertain. The findings of this trial will provide evidence-based guidance on graft material selection in extraction site management. If one graft type proves superior, this would validate the use of donated human teeth as a sustainable and effective bone graft source, potentially reducing reliance on animal-derived or synthetic substitutes. Ultimately, optimizing socket grafting methods is expected to enhance outcomes in implant and prosthetic dentistry by preserving bone anatomy and facilitating successful restorative treatments.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 60 years.

Medically healthy patients classified as ASA I.

Presence of a single non-restorable tooth indicated for extraction in the posterior maxilla.

Adequate oral hygiene, with plaque and bleeding indices both below 20%.

Sufficient bone volume to allow socket preservation without requiring simultaneous augmentation.

Patients willing to participate in the study and able to provide written informed consent.

Ability to commit to follow-up visits for up to 6 months.

Exclusion Criteria:

Smokers or tobacco users of any form.

Presence of uncontrolled systemic diseases (e.g., uncontrolled diabetes).

Conditions affecting bone metabolism (e.g., osteoporosis, long-term corticosteroid therapy).

Pregnant or lactating women.

History of radiotherapy in the head and neck region.

Active infection or suppuration at the extraction site.

Immunocompromised patients or those on immunosuppressive therapy.

Patients taking medications known to impair healing (e.g., bisphosphonates).

Allergy or hypersensitivity to any study-related materials.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Alveolar Ridge Width (Buccolingual Dimension) | Baseline (immediately after extraction) and 6 months post-operative
  Measurement of the buccolingual width of the alveolar ridge using standardized Cone-Beam Computed Tomography (CBCT). Width is measured at predetermined reference points to assess dimensional bone changes following grafting.
Change in Alveolar Ridge Height (Vertical Dimension) | Baseline and 6 months post-operative
  Vertical height of the alveolar ridge measured radiographically on CBCT at standardized anatomical landmarks to quantify bone height changes over the healing period.
Bone Density at the Grafted Site | 6 months post-operative
  Bone density at the extraction site measured using CBCT expressed in Hounsfield Units (HU) to evaluate bone quality gained after grafting

SECONDARY OUTCOMES:
Postoperative Pain Levels (VAS Score) | 24, 48, and 72 hours post-operative
  Postoperative pain will be evaluated using a Visual Analog Scale (VAS) ranging from 0 to 10, where 0 indicates no pain and 10 indicates severe pain. Participants will record pain levels at predefined postoperative intervals.
Postoperative swelling | Baseline (preoperative), 24, 48, and 72 hours post-operative
  Facial swelling will be assessed through standardized digital facial photographs taken at each time point. Facial dimensions will be analyzed using image analysis software to quantify postoperative edema.
Patient Satisfaction Score | 6 months post-operative
  Patient satisfaction will be recorded using a structured questionnaire that scores satisfaction on a scale from 0 to 4 (0 = very satisfied, 4 = very dissatisfied). Participants will complete the questionnaire at designated follow-up intervals.
Width of Keratinized Tissue | Baseline and 6 months post-operative
  Keratinized tissue width will be measured using a UNC-15 periodontal probe at the buccal aspect of the site. Measurements will be taken at baseline and during the final follow-up to assess changes associated with socket healing.
Histomorphometric Analysis of Bone Core Biopsies | 6 months post-operative (at implant placement)
  Histological assessment of bone core biopsies harvested at implant placement will determine the percentage of newly formed bone, residual graft particles, and connective tissue within the specimen using calibrated image analysis software

CONTACTS AND LOCATIONS:
Overall Officials: Enas Elgendy, PhD, Study Chair — Faculty of Dentistry, Kafrelsheikh University; Ahmed Elgendy, PhD, Principal Investigator — Faculty of Dentistry, Kafrelsheikh University; Abir El-Mouelhy, PhD, Principal Investigator — National Research Centre, Cairo, Egypt
Locations (1):
- Faculty of Dentistry, Kafrelsheikh University, Kafr ash Shaykh, Egypt